CLINICAL TRIAL: NCT02213354
Title: A Phase II Randomized, Partially-Blinded, Controlled Trial in Healthy Adults Aged 65 Years and Older to Assess the Safety, Reactogenicity, and Immunogenicity of an MF59-Adjuvanted, Monovalent Inactivated Influenza A/H7N9 Virus Vaccine Administered Intramuscularly at Different Intervals and Dosages
Brief Title: H7N9 Mix and Match With MF59 in Healthy Elderly Persons
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 13-0034; HHSN272201300016I
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2016-04

CONDITIONS: Avian Influenza
Keywords: Influenza, H7N9, Elderly, Vaccine, MF59 Adjuvant
MeSH Terms: conditions — Influenza in Birds; Influenza, Human | interventions — MF59 oil emulsion; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Group 2 (Experimental): 60 subjects receive Sanofi A/H7N9 antigen 3.75 mcg plus Novartis MF59 adjuvant IM on Day 1, Day 57, and Day 169
  Interventions: Drug: MF59; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group 6 (Experimental): 60 subjects receive Sanofi A/H7N9 antigen 15 mcg plus Novartis MF59 adjuvant IM on Day 1, Day 57, and Day 169
  Interventions: Drug: MF59; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group 5 (Experimental): 60 subjects receive Sanofi A/H7N9 antigen 15 mcg plus Novartis MF59 adjuvant IM on Day 1, Day 29 and Day 169
  Interventions: Drug: MF59; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group 4 (Experimental): 60 subjects receive Sanofi A/H7N9 antigen 7.5 mcg plus Novartis MF59 adjuvant IM on Day 1, Day 57, and Day 169
  Interventions: Drug: MF59; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group I (Experimental): 60 subjects receive Sanofi A/H7N9 antigen 3.75 mcg plus Novartis MF59 adjuvant intramuscularly (IM) on Day 1, Day 29 and Day 169
  Interventions: Drug: MF59; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013
- Group 3 (Experimental): 60 subjects receive Sanofi A/H7N9 antigen 7.5 mcg plus Novartis MF59 adjuvant IM on Day 1, Day 29 and Day 169
  Interventions: Drug: MF59; Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013

INTERVENTIONS:
Drug: MF59 — Microfluoridized adjuvant 59 (MF59) is an oil-in-water emulsion. Group 1-6 receive 3.75 mcg, 7.5 mcg and 15 mcg.
Biological: Influenza Virus Vaccine, Monovalent A/H7N9 A/Shanghai/2/2013 — Monovalent inactivated split influenza virus vaccine made with HA antigen derived from the influenza A/Shanghai/2/2013 virus. Monovalent influenza A/H7N9 virus vaccine. Group 1-6 receive 3.75 mcg, 7.5 mcg and 15 mcg.

SUMMARY:
This is a Phase II randomized, partially-blinded, controlled trial in 360 (up to 600) males and females, 65 years of age and older, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of a monovalent inactivated influenza A/H7N9 virus vaccine manufactured by Sanofi Pasteur administered intramuscularly at different intervals and dosages (3.75, 7.5, or 15 mcg of HA/0.5 mL dose) given with MF59 adjuvant manufactured by Novartis Vaccines and Diagnostics. Subjects will receive three doses of the vaccine. Safety, reactogenicity, and immunogenicity data will be collected at standard time points with safety follow-up to continue through one year post dose 2. Study Duration is approximately 30 months and Subject Participation is approximately 18 months. The primary objectives are to (1) assess the safety and reactogenicity of different dosages (3.75, 7.5, and 15 mcg of HA/0.5 mL dose) of an MF59-adjuv

DETAILED DESCRIPTION:
This is a Phase II randomized, partially-blinded, controlled trial in males and females, 65 years of age and older, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of a monovalent inactivated influenza A/H7N9 virus vaccine, derived from the influenza A/Shanghai/2/2013 virus, manufactured by Sanofi Pasteur administered intramuscularly at different intervals and dosages (3.75, 7.5, or 15 mcg of HA/0.5 mL dose) given with MF59 adjuvant manufactured by Novartis Vaccines and Diagnostics. Subjects will be assigned randomly to 1 of 6 groups (60 to 100 subjects per group) to receive three doses intramuscularly of the inactivated A/H7N9 vaccine at dosages (3.75, 7.5, or 15 mcg of HA/0.5 mL dose) given with MF59 adjuvant using two different study vaccination schedules. The first and third study vaccinations will be administered to all subjects on Day 1 and approximately Day 169. The second study vaccination will be administered either on approximately Day 29 for Groups 1, 3, and 5 or approximately Day 57 for Groups 2, 4, and 6. Reactogenicity will be measured from the time of each study vaccination through 8 days after each study vaccination by the occurrence of solicited injection site and systemic reactions. Unsolicited non-serious adverse events (AEs) will be collected from the time of each study vaccination through approximately 28 days after each study vaccination. Serious adverse events (SAEs) and new-onset chronic medical conditions will be collected from the time of the first study vaccination through approximately 12 months after the last study vaccination.

Immunogenicity testing will include performing hemagglutination inhibition (HAI) and neutralizing (Neut) antibody assays on serum obtained immediately prior to the first study vaccination (Day 1), approximately 28 days after the second study vaccination (approximately Day 57 for Groups 1, 3, and 5; approximately Day 85 for Groups 2, 4, and 6), immediately prior to the third study vaccination (approximately Day 169), and approximately 28 days after the third study vaccination (approximately Day 197). Subjects in Groups 1, 3, and 5 will also have immunogenicity testing for HAI and Neut antibody assays performed on serum obtained at approximately 56 days after the second study vaccination (approximately Day 85). Between 360 and 600 subjects will be enrolled in this trial. Study Duration is approximately 30 months and Subject Participation is approximately 18 months. The primary objectives are to (1) assess the safety and reactogenicity of different dosages (3.75, 7.5, and 15 mcg of HA/0.5 mL dose) of an MF59-adjuvanted, monovalent inactivated influenza A/H7N9 virus vaccine using two different study vaccination schedules and (2) assess the serum hemagglutination inhibition (HAI) antibody responses to different dosages (3.75, 7.5, and 15 mcg of HA/0.5 mL dose) of an MF59-adjuvanted, monovalent inactivated influenza A/H7N9 virus vaccine using two different study vaccination schedules following receipt of the second study vaccination. The secondary obectives are to (1) assess study vaccine-related unsolicited non-serious adverse events following receipt of different dosages (3.75, 7.5, and 15 mcg of HA/0.5 mL dose) of an MF59-adjuvanted, monovalent inactivated influenza A/H7N9 virus vaccine using two different study vaccination schedules, (2) assess new-onset chronic medical conditions following receipt of different dosages (3.75, 7.5, and 15 mcg of HA/0.5 mL dose) of an MF59-adjuvanted, monovalent inactivated influenza A/H7N9 virus vaccine using two different study vaccination sched

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Are males or females, 65 years of age and older.
4. Are in good health1. 1As determined by medical history and targeted physical examination, if indicated based on medical history, to evaluate acute or currently ongoing chronic medical diagnoses or conditions that would affect the assessment of eligibility and safety of subjects. Chronic medical diagnoses or conditions being actively managed must be within acceptable limits in the last 180 days. Good health in the elderly is also defined as no change in chronic prescription medication, dose, or frequency of medication in the 90 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and does not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and first study vaccination are acceptable provided the subject is asymptomatic, condition stable, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Topical, nasal, and inhaled medications (with the exception of steroids as outlined in the Subject Exclusion Criteria (see Section 5.2)), herbals, vitamins, and supplements are permitted
5. Oral temperature is less than 100.0 degrees F.
6. Pulse is 50 to 115 bpm, inclusive.
7. Systolic blood pressure is 85 to 160 mm Hg, inclusive.
8. Diastolic blood pressure is 55 to 95 mm Hg, inclusive

Exclusion Criteria:

1. Have an acute illness2, as determined by the site principal investigator or appropriate sub-investigator, within 72 hours prior to study vaccination.

2An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.

2. Have any medical disease or condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation3.

3Including acute or chronic medical disease or condition, defined as persisting 3 months (defined as 90 days) or longer, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this study.

3. Reside in a nursing home4 or other skilled nursing facility or have a requirement for skilled nursing care.

4An ambulatory subject who does not require skilled nursing care and is a resident of a retirement home or community is eligible for this clinical trial.

4. Inability to provide informed consent or complete study activities, for example, due to dementia or other impairment.

5. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.

6. Have known active neoplastic disease or a history of any hematologic malignancy.

7. Have known HIV, hepatitis B, or hepatitis C infection. 8. Have known hypersensitivity or allergy to eggs, egg or chicken protein, squalene-based adjuvants, or other components of the study vaccine.

9. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines.

10. Have a history of Guillain-Barré Syndrome. 11. Have a history of neuralgia, paresthesia, neuritis, convulsions, or encephalomyelitis within 90 days prior to study vaccination.

12. Have a history of autoimmune disease5. 5Including, but not limited to, autoimmune processes resulting in neuroinflammatory diseases, vasculitis, clotting disorders, dermatitis, arthritis, thyroiditis, or muscle, liver, or kidney disease.

13. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.

14. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.

15. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.

16. Have taken oral or parenteral corticosteroids of any dose within 30 days prior to study vaccination.

17. Have taken high-dose inhaled corticosteroidswithin 30 days prior to study vaccination. High-dose defined as >800 mcg/day of beclomethasone dipropionate CFC or equivalent.

18. Received a licensed live vaccine within 30 days prior to enrollment in this study, or plans to receive a licensed live vaccine within 30 days before or after each study vaccine.

19. Received a licensed inactivated vaccine within 14 days prior to enrollment in this study, or plans to receive a licensed inactivated vaccine within 14 days before or after each study vaccine.

20. Received immunoglobulin or other blood products within 90 days prior to study vaccination.

21. Received an experimental agent6 within 30 days prior to the first study vaccination, or expects to receive an experimental agent7 during the 18-month study period.

6Including vaccine, drug, biologic, device, blood product, or medication. 7Other than from participation in this study. 22. Are participating or plan to participate in another clinical trial with an interventional agent8 during the 18-month study period.

8 Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.

23. Prior participation in a clinical trial of influenza A/H7 vaccine9 or have a history of A/H7 actual or potential exposure or infection prior to the first study vaccination.

9And assigned to a group receiving influenza A/H7 vaccine, does not apply to documented placebo recipients.

24. Plan to travel outside the US (continental US, Hawaii, and Alaska) within the 28 days following each study vaccination.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 479 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the A/H7N9 antigen contained in the study vaccine | 28 days after the second study vaccination
Percent of subjects achieving HAI seroconversion against the A/H7N9 antigen contained in the study vaccine (either a pre-vaccine HAI titer < 1:10 and a post-vaccine HAI titer > /= 1:40 or a pre-vaccine HAI titer > /=1:10 and a min 4-fold rise in post-vac | 28 days after the second study vaccination
Occurrence of study vaccine-related serious adverse events | Through Day 1 to 12 months after the last study vaccination
Occurrence of solicited injection site and systemic reactogenicity events | Through 8 days after each study vaccination

SECONDARY OUTCOMES:
Occurrence of study vaccine-related unsolicited non-serious adverse events | 28 days after each study vaccination
Occurrence of new-onset chronic medical conditions | Through Day 1 to 12 months after the last study vaccination
Percentage of subjects achieving Neut seroconversion against A/H7N9 antigen (either prevaccination Neut titer < 1:10 and postvaccination Neut titer > /=1:40 or prevaccination Neut titer > /=1:10 and minimum fourfold rise in post-vaccination Neut | 28 days after the second and third study vaccinations
Geometric Mean Titers of serum HAI and Neut antibodies against the A/H7N9 antigen | Baseline and 28 days after the second and third study vaccinations
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the A/H7N9 antigen contained in the study vaccine | Baseline and 28 days after the third study vaccination
Percentage of subjects achieving a serum Neut antibody titer of 1:40 or greater against the A/H7N9 antigen contained in the study vaccine | Baseline and 28 days after the second and third study vaccinations
Percentage of subjects achieving HAI seroconversion against the A/H7N9 antigen | 28 days after the third study vaccination

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Duke Human Vaccine Institute - Duke Clinical Vaccine Unit, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Vanderbilt University Medical Center - Vanderbilt Institute for Clinical and Translational Research - Clinical Research Center (VICTR-CRC), Nashville, Tennessee
  - University of Texas Medical Branch - Sealy Center for Vaccine Development - Clinical Trials Group, Galveston, Texas
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Group Health Research Institute - Seattle - Vaccines and Infectious Diseases, Seattle, Washington